CLINICAL TRIAL: NCT02287753
Title: Relationship Between Parameters of Vascular Occlusion Test Using Near Infrared Spectroscopy and Clinical Parameters & Outcomes in Pediatric Cardiac Surgery
Brief Title: Relationship Between Parameters of VOT Using NIRS and Clinical Outcomes in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-1309-095-522
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Congenital Heart Disease
Keywords: vascular occlusion test; near infrared spectroscopy
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vascular occlusion test (VOT) (Experimental): Pediatric patients aged under 8 years old are enrolled in this study. VOT is performed in 3 times : after induction of anesthesia, during cardiopulmonary bypass (CPB) for main surgical procedure and after weaning from CPB. The relationship between postoperative outcome variables and the dynamic parameters from VOT, such as desaturation and reoxygenation rate, and reactive hyperemic area, will be evaluated.
  Interventions: Other: vascular occlusion test using Pediatric SomaSensor for INVOS 5100C

INTERVENTIONS:
Other: vascular occlusion test using Pediatric SomaSensor for INVOS 5100C — Pediatric SomaSensor for INVOS 5100C is attached at calf muscle and non-invasive blood pressure cuff is applied to ipsilateral thigh. VOT is performed as: after baseline oxygen saturation value is recorded, cuff pressure is rapidly increased to 30 mmHg over than systolic blood pressure. After 3 minutes of ischemic time, cuff pressure is rapidly decreased. It is performed at 3 time periods : before start of operation, during cardiopulmonary bypass, and after weaning from cardiopulmonary bypass.

SUMMARY:
The purpose of this study is to evaluate the ability of vascular occlusion test (VOT) during cardiac surgery to predict postoperative outcomes in pediatric patients.

DETAILED DESCRIPTION:
After induction of anesthesia, pediatric SomaSensor for INVOS 5100C is attached at calf muscle and non-invasive blood pressure cuff is applied to ipsilateral thigh. VOT is performed as: after baseline oxygen saturation value is recorded, cuff pressure is rapidly increased to 30 mmHg over than systolic blood pressure. After 3 minutes of ischemic time, cuff pressure is rapidly decreased. It is performed at 3 time periods : before start of operation, during cardiopulmonary bypass, and after weaning from cardiopulmonary bypass. Postoperative outcome variables are recorded after surgery : major adverse event, use of inotropic and vasoactive drugs, duration of mechanical ventilation and ICU stay. The relationship between the results of VOT and postoperative outcome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged under 8 years old who are scheduled for cardiac surgery

Exclusion Criteria:

* Skin disease
* Skin preparation involving thigh
* Peripheral vascular disease

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Major adverse event | up to 1 years after surgery
  Major adverse event is defined as cardiac compression, re-sternotomy because of hemodynamic instability, ECMO support, Cr> 2mg/dL, cerebral hemorrhage or infarct and mortality.

SECONDARY OUTCOMES:
Use of inotropic and vasoactive drugs | up to 1 years after surgery
  Use of inotropic and vasoactive drugs is evaluated using vasoactive-Inotropic scores (VIS). VIS is calculated as: dopamine dose (㎍/kg/min) + dobutamine dose (㎍/kg/min) + 100 x epinephrine dose (㎍/kg/min) + 10 x milrinone dose (㎍/kg/min) + 10,000 x vasopressin dose (U/kg/min) + 100 x norepinephrine dose (㎍/kg/min).(7) VIS at 0, 24, 48, and 72 hours after surgery ended are collected in all patients.
Length of mechanical ventilation time and ICU stay | up to 1 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Jang YE, Song IK, Kim EH, Kim HS, Kim JT. Near-Infrared Spectroscopy and Vascular Occlusion Test for Predicting Clinical Outcome in Pediatric Cardiac Patients: A Prospective Observational Study. Pediatr Crit Care Med. 2018 Jan;19(1):32-39. doi: 10.1097/PCC.0000000000001386. PMID 29140967